CLINICAL TRIAL: NCT00740285
Title: Effectiveness and Safety of Lidocaine for Scleroderma. Randomized Double-Blind Clinical Trial
Brief Title: Effectiveness and Safety of Lidocaine for Scleroderma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 390/00
Record Dates: First submitted 2008-08-19; First posted 2008-08-22 (Estimated); Last update posted 2008-08-22 (Estimated); Status verified 2008-08

CONDITIONS: Scleroderma
Keywords: scleroderma; scleroderma - limited or diffuse types; lidocaine; effectiveness
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Limited | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Lidocaine 2% without vessel constrictor
- 2 (Placebo Comparator)
  Interventions: Other: Placebo - physiological solution 0,9%

INTERVENTIONS:
Drug: Lidocaine 2% without vessel constrictor — * first 5 days: 20ml lidocaine 2% without vessel constrictor + physiological solution 0,9% 500ml intravenously during 4 hours
  * next 5 days: 30ml lidocaine 2% without vessel constrictor + physiological solution 0,9% 500ml intravenously during 4 hours total: 10 days
  Arms: 1
Other: Placebo - physiological solution 0,9% — first 5 days: 20ml of physiological solution 0,9% 500ml + physiological solution 0,9% 500ml intravenously during 4 hours next 5 days: 30ml of physiological solution 0,9% 500ml + physiological solution 0,9% 500ml intravenously during 4 hours total: 10 days
  Arms: 2

SUMMARY:
Scleroderma, or systemic sclerosis, is a chronic connective tissue disease generally classified as one of the autoimmune rheumatic diseases. The disease is characterized by thickening and fibrosis skin, affecting vessels and many organs such as the esophagus, stomach, bowls, lung, heart and kidney. The exact cause or causes of scleroderma are still unknown, but scientists and medical investigators in a wide variety of fields are working hard to make those determinations. It is known that scleroderma involves overproduction of collagen.

FLICKMAN et al, in 1973 published an article about the role of lidocaine at prolyl-hydroxylase activity decrease, which is an important enzyme of collagen production. Until now, there is only a case series showing the improvement of thickening skin (75%) and esophagus symptoms (66%) after intravenous lidocaine 2% during 10 days. So it is necessary a RCT to prove these findings.

ELIGIBILITY:
Inclusion Criteria:

* Scleroderma (diffuse or limited) at less than 5 years of the first symptom

Exclusion Criteria:

* Overlap with other connective tissue diseases
* Fibromyalgia
* Pregnancy
* Current use of ciclofosfamide ou D-penicillamine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-04; Primary Completion 2006-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Skin thickening evaluated by Skin Score | before, immediately after the intervention and 6 months later

SECONDARY OUTCOMES:
Safety - evaluated by the adverse effects during the intervention | immediately after the intervention
Quality of Life evaluated by HAQ | before, immediately after the intervention and 6 months later
Pressure at lower esophagus evaluated by esophagus manometry | before, immediately after the intervention and 6 months later
Vessel alterations (as the number deletion/ectasia) evaluated by fingernail capillaroscopy | before, immediately after the intervention and 6 months later
Subjective evaluation by patients | before, immediately after the intervention and 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Riera, MD, Principal Investigator — Universidade Federal de São Paulo; Virginia FM Trevisani, PhD, Study Chair — Universidade Federal de São Paulo; Alexandre WS Silva, PhD, Study Director — Universidade Federal de São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Jimenez SA, Hitraya E, Varga J. Pathogenesis of scleroderma. Collagen. Rheum Dis Clin North Am. 1996 Nov;22(4):647-74. doi: 10.1016/s0889-857x(05)70294-5. PMID 8923589